CLINICAL TRIAL: NCT06339931
Title: Effects of Lumber Spine Mobilization, Leg Movement, and Spinal Traction With and Without Belt in Patients With Lumber Radiculopathy.
Brief Title: Lumber Spine Mobilization and Spinal Traction on Lumber Radiculopathy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR &AHS/23/0181
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Lumbar Radiculopathy
Keywords: Lumber Radiculopathy; Low Back Pain; Quality of Life; Traction
MeSH Terms: conditions — Radiculopathy; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMWLM combined Spinal traction with belt (Experimental): Group A (Spinal traction with belt plus SMWLM) as per Mulligan rule of three SMWLM on affected lumbar vertebrae. Spinal traction with belt for 10 mins.
  Interventions: Other: SMWLM combined Spinal traction with belt
- SMWLM combined Spinal traction without belt (Active Comparator): Group B (Spinal traction without belt plus SMWLM) as per Mulligan rule of three SMWLM on affected lumbar vertebrae. Manual spinal traction technique without belt.
  Interventions: Other: SMWLM combined spinal traction without belt

INTERVENTIONS:
Other: SMWLM combined Spinal traction with belt — Group A, therapist 1 will stand at the participant's ventral side and apply a transverse glide with the thumb on the involved lumbar spinous process. Therapist 2 will then abduct the affected leg by 10° and take the limb gently into hip flexion with the knee extended, while the glide will be sustained continuously by Therapist. Wrap the traction belt around both your hips and the proximal aspect of the patient's thighs.Apply traction by leaning backward and shifting your body weight onto your posterior leg.
  Arms: SMWLM combined Spinal traction with belt
Other: SMWLM combined spinal traction without belt — Group B, therapist 1 will stand at the participant's ventral side and apply a transverse glide with the thumb on the involved lumbar spinous process. Therapist 2 will then abduct the affected leg by 10° and take the limb gently into hip flexion with the knee extended, while the glide will be sustained continuously by Therapist. Manual traction is applied by placing the patient over a rolled pillow while lying sideways. The roll should be 6-8 inches in diameter and should be placed at the level of the spine where the traction or separation is to occur. Pull the patient's legs toward you as you lean your body backward to apply a traction force.
  Arms: SMWLM combined Spinal traction without belt

SUMMARY:
Lumber radiculopathy, also known as sciatica, is a condition that causes pain in the lower back and legs due to irritation or compression of the spinal nerves. group between 20 and 50 years old. This study will explore the effects of lumbar spine mobilization with leg movement and spinal traction with and without belt in patients with pain and functional limitations due to lumbar radiculopathy. A randomized control trial will be conducted at Atta Jaspal Hospital and Trauma Center through convenient sampling technique on 44 patients, which will be allocated through simple random sampling through sealed opaque envelopes into groups A and B. Group A will be treated with SMWLM, conventional electrotherapy, and traction without a belt, and Group B will be treated with SMWL, conventional electrotherapy, and lumbar traction with a belt. A pretreatment baseline will be set for pain, ROM, and disability at the lumbar spine by using the NPRS, inclinometer, and ODI questioner. Follow-up will be conducted after 4 weeks of post-treatment sessions. The intensity of pain, range of motion, and disability index will be evaluated using the NPRS, inclinometer, and ODI questionnaire. The data will be analyzed using SPSS software version 26. The conclusion of the study will be based on either accepting or rejecting the null and alternate hypotheses.

DETAILED DESCRIPTION:
Low back pain (LBP) is one of the primary causes of disability worldwide. Most people-between 50% and 80%-experience LBP at some point in their life. It limits the ability to perform daily activities, such as walking, standing, or lifting objects. It can also lead to decreased mobility, reduced work productivity, and increased healthcare costs. Radiating pain is commonly caused by lumbar intervertebral disk abnormalities, which are linked with nerve root irritation and affect 3% to 10% of people with generalized low back pain. Sciatica, another name for lumbar radiculopathy, is a disorder marked by pain, weakness, numbness, or tingling sensations that radiate down the lower back along a nerve root, frequently into the buttock, thigh, and lower leg. One or more lumbar nerve roots are usually compressed, irritated, or inflamed as a reason.

ELIGIBILITY:
Inclusion Criteria:

* Age of 16-50 years of both sexes, unilateral radiculopathy in the distribution of specific nerve with positive straight leg raise (SLR).
* Mild to moderate disability and pain on a scale of NPRS < 7, minimum chronicity of 1 month, and maximum 6 months

Exclusion Criteria:

* Patients with previous spinal surgery'
* Any bony or soft tissue systemic disease.
* Patients with diagnosed case of co morbidities such as malignancies , RA or fractures that causes bilateral leg pain

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | 4 weeks
  The NPRS scale will be used to quantify pain intensity levels. The scale ranges from '0' for the least amount of pain ("no pain") to '10' for the most extreme levels of pain ("pain as severe as you can imagine")
Inclinometer | 4 weeks
  Bubble inclinometer for measuring joint range of motion
Oswestry Disability Index | 4 weeks
  Gold standard of low back pain functional outcome tools

CONTACTS AND LOCATIONS:
Overall Officials: Shakil Ur Rehman, Principal Investigator — Riphah International University
Locations (1):
- Atta Jaspal Hospital and ortho trauma center, Bhalwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No